CLINICAL TRIAL: NCT05339776
Title: Evaluation of Hand Lateralization Cognitive Task From Different Personal Perspectives by Using EEG Analysis Method in Amputees
Brief Title: Hand Lateralization by Using EEG Analysis Method in Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Burcu Dilek, PhD, Principal Investigator, Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6568
Record Dates: First submitted 2022-04-01; First posted 2022-04-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Body Image
Keywords: EEG; mental rotation; hand lateralization; hand recognition; amputees; body schema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One of groups: amputees group (Active Comparator): We planned to enroll two groups to the study. One group is named "amputees" the other one is "control". Both groups will enroll "hand lateralization" for at least 10 days. Before and after comparisons will be analyzed.
  Interventions: Behavioral: Hand Lateralization Test
- One of groups: control group (Active Comparator): Control group will be matched in terms of age and gender with the amputees group.
  Interventions: Behavioral: Hand Lateralization Test

INTERVENTIONS:
Behavioral: Hand Lateralization Test — Before hand lateralization test, participants will be evaluated. Both groups (Amputees and Control) will complete hand lateralization test for at least 10 days. The test will be sent each day on an online system. Participants' performances will be recorded via online system. After hand lateralization test, participants will be evaluated.

SUMMARY:
Studies on the improvement of body image or body perception have proven their effectiveness in different clinical situations such as pain management and chronic pain treatment. The aim of this study is to evaluate the hand lateralization cognitive task by recording Electroencephalography (EEG) signals from different personal perspectives in amputees. In this study, the paradigm in which personal perspectives are evaluated over the hand lateralization task will be applied to amputees and healthy volunteer participants. Data will be recorded via EEG and Eprime software program.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the hand lateralization cognitive task by recording Electroencephalography (EEG) signals from different personal perspectives in amputees.

In this study, the paradigm in which personal perspectives are evaluated over the hand lateralization task will be applied to amputees and healthy volunteer participants.

It was planned to enroll two groups to the study. One group is named "amputees" the other one is "control". Control group will be matched in terms of age and gender with the amputees group. Before hand lateralization test, participants will be evaluated regarding eligible criterias and EEG paradigm regarding hand lateralization will be performed for each participant.

Both groups (Amputees and Control) will complete "hand lateralization program" for at least 10 days. The test will be sent each day on an online system. Participants' performances will be recorded via online system.

Following 10-day period, EEG paradigm regarding hand lateralization will be performed for each participant, again.

Before and after comparisons will be analyzed. Data will be recorded via EEG and Eprime software program.

EEG-Event Related Oscillation (power spectrum, phase locking) analysis will be performed for each frequency bands: alpha, theta, beta, gamma.

Eprime analysis will be performed for the data of reaction time and accuracy rate.

ELIGIBILITY:
Control group:

Inclusion Criteria:

* being between ages 18-65,
* consenting,
* with no limitation in mobility or movement disorder,
* A score of 21 or higher on the Montreal Cognitive Assessment Test

Exclusion Criteria:

* refuse to attend to the study,
* Having any mental, neurological or musculoskeletal problems,
* Inability to perform activities that require long-term attention,
* Inability to detect given commands,
* Using sedative drugs and/or derivatives

Amputee group:

Inclusion Criteria:

* between ages 18-65,
* using prosthesis,
* A score of 21 or higher on the Montreal Cognitive Assessment Test

Exclusion Criteria:

* Having phantom pain,
* Having open wound on stump,
* Having any discomfort feeling on stump,
* Having any mental, neurological or musculoskeletal problems,
* Inability to perform activities that require long-term attention,
* Inability to detect given commands,
* Using sedative drugs and/or derivatives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) frequency bands: alpha, theta, beta, gamma | Before and after the hand lateralization test: 10-14 days
  Changes in power spectrum and phase locking

SECONDARY OUTCOMES:
Reaction time to decide whether the hand is right or left | Before and after the hand lateralization test: 10-14 days
  E-prime parameter: recorded as milisecond
Accuracy proportion of given answers regarding hand lateralization | Before and after the hand lateralization test: 10-14 days
  E-prime parameter: recorded as percentage

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Dilek, PhD, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No